CLINICAL TRIAL: NCT00653575
Title: HIV Risk Among Women With a History of Childhood Sexual Abuse
Brief Title: Adult Sexual Risk Behavior Among Women With a History of Childhood Sexual Abuse
Status: Completed | Type: Observational
Sponsor: Syracuse University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Theresa E. Senn, PhD, Syracuse University
Other Study IDs: R21MH083502 (NIH); R21MH083502 (NIH); DAHBR 9A-ASPQ
Record Dates: First submitted 2008-04-03; First posted 2008-04-07 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: HIV Infections; Child Abuse, Sexual
Keywords: Sexual Behavior; HIV; Sexually Transmitted Diseases
MeSH Terms: conditions — HIV Infections; Coitus; Sexual Behavior; Sexually Transmitted Diseases | interventions — Information Motivation Behavioral Skills Model

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Women who report a history of childhood sexual abuse
  Interventions: Behavioral: Information-Motivation-Behavioral Skills model; Behavioral: Traumagenic Dynamics model
- 2: Women who do not report a history of childhood sexual abuse
  Interventions: Behavioral: Information-Motivation-Behavioral Skills model; Behavioral: Traumagenic Dynamics model

INTERVENTIONS:
Behavioral: Information-Motivation-Behavioral Skills model — The Information-Motivation-Behavioral Skills model is an influential and empirically supported theory of health behavior. The model suggests that HIV-related information, motivation, and behavioral skills are important determinants of sexual behavior; thus, childhood sexual abuse may lead to deficits in these areas. This model will be used to guide research interviews.
Behavioral: Traumagenic Dynamics model — The Traumagenic Dynamics model is an influential and empirically supported model of the effects of childhood sexual abuse. The model suggests that childhood sexual abuse leads to traumatic sexualization, stigmatization, betrayal, and powerlessness and that these four traumagenic dynamics lead to adverse outcomes, including increased rates of sexual risk behavior. This model will be used to guide research interviews.

SUMMARY:
This study will evaluate whether childhood experiences are related to current sexual behavior of adult women.

DETAILED DESCRIPTION:
Adverse childhood events, including physical and sexual abuse, can cause significant distress for those affected, during both childhood and adulthood. Childhood abuse appears to increase the risk of a number of negative outcomes later in life, including psychiatric disorders, substance abuse, and HIV and sexually transmitted infections. Previous research has consistently found an association between childhood sexual abuse and greater rates of adult sexual risk behavior. However, improved understanding of how childhood sexual abuse relates to adult sexual risk behavior is needed. The Information-Motivation-Behavioral Skills and Traumagenic Dynamics models are theories used to investigate determinants of sexual behavior and effects of childhood abuse. Using these models to examine the relationship between childhood sexual abuse and adult sexual risk behavior may help in creating effective sexual risk reduction interventions for women abused during childhood. This study will evaluate whether childhood experiences are related to current sexual behavior of adult women. The study will also evaluate which theory, the Information-Motivation-Behavioral Skills model or the Traumagenic Dynamics model, better mediates the relationship between childhood sexual abuse and adult sexual risk behavior.

Participation in this study will include one study visit. Participants will first complete a 45-minute computerized survey that includes questions about childhood experiences; family environment; current health and behavior; attitudes, knowledge, and thoughts about sex and relationships; control over life circumstances; and substance use. Participants will then engage in two brief role plays in which they will either make a request of their partner or must stand up for themselves. For the last part of the visit, participants will be asked questions about condoms and condom use and will be asked to place a condom on a model used in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Understands English

Exclusion Criteria:

* Impaired mentally

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include women seeking treatment at the Monroe County Health Department STD Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 481 (Actual)
Dates: Start 2008-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Number of sexual partners | Measured at Month 3

SECONDARY OUTCOMES:
Frequency of unprotected intercourse | Measured at Month 3
Proportion of episodes of unprotected intercourse | Measured at Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Theresa E. Senn, PhD, Principal Investigator — Syracuse University
Locations (1):
- Monroe County Health Department STD Clinic, Rochester, New York, United States